CLINICAL TRIAL: NCT02298764
Title: Somatic Experiencing for Patients With Comorbid Posttraumatic Stress and Back Pain - A Randomized Controlled Trial.
Brief Title: Back Pain and PostTraumaticStressDisorder. A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Spine Centre of Southern Denmark (Other)
Responsible Party: Principal Investigator, Tonny Elmose Andersen, phd., associate professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT2014PTSD
Record Dates: First submitted 2014-11-12; First posted 2014-11-24 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Low Back Pain; PTSD
MeSH Terms: conditions — Low Back Pain; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard + 10 psychotherapeutic sessions (Active Comparator): - standard back pain treatment plus 10 psychotherapeutic sessions, that will include the shock-trauma method 'Somatic Experiencing'.
  Interventions: Other: Standard back pain treatment + 10 psychotherapeutic sessions
- Standard back pain treatment (Active Comparator): Standard back pain treatment
  Interventions: Other: Standard back pain treatment

INTERVENTIONS:
Other: Standard back pain treatment — Standard back pain treatment
  Arms: Standard back pain treatment
Other: Standard back pain treatment + 10 psychotherapeutic sessions — Standard back pain treatment plus 10 psychotherapeutic session, that will include the shock-trauma method "somatic experiencing".
  Arms: standard + 10 psychotherapeutic sessions

SUMMARY:
Aim The aim is to test whether a short psychotherapeutic intervention targeting Post Traumatic Stress Disorder (PTSD) symptoms will have an additional positive effect on the outcomes of the Standard Multidisciplinary Program (SMP) against chronic back pain development.

DETAILED DESCRIPTION:
Focus Patients with back pain often demonstrate symptoms of PTSD measured via the Harvard Trauma Questionnaire Scale (HTQ). It has been found that PTSD and pain may maintain each other.

Methods Thousand consecutive patients with Low Back Pain (LBP) referred to the Spine Center are screened for PTSD. It is expected that 100 patients will meet the inclusion criteria and be randomized to SMP or to SMP plus 10 psychotherapeutic sessions, that will include the shock-trauma method 'Somatic Experiencing'.

Conclusion The project started in 2013, so there have not yet been any results. Currently total reached 65 back pain patients; 34 patients in the SMP + sessions intervention arm.

Effect parameters are: Pain, daily function, EuroQOL and (HTQ), anxiety and depression, fear avoidance (Tampa Scale for Kinesiophobia) on entry, and at 6/12 months.

This "Nested Randomized Trial in a Cohort Design" is one of the very first studies targeting both PTSD and chronic pain-related symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Back pain: from 1/2 Y duration or longer
* Trauma according to HTQ

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Functional status, Roland Morris Scale | 0, 1 year
  scale ranging from 0-24

SECONDARY OUTCOMES:
Harvard Trauma Questionnaire | 0, 1 year
  scale ranging from 17-68
Back pain intensity, numeric rating scale | 0, 1 year
  scale ranging from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Tonny E Andersen, PhD, Principal Investigator — University of Southern Denmark, Department of Psychology
Locations (1):
- University of Southern Denmark, Odense, Fyn, Denmark